CLINICAL TRIAL: NCT03238326
Title: A Long-term, Multicenter, Open-label Trial to Evaluate the Safety and Tolerability of Flexible-Dose Brexpiprazole as Maintenance Treatment in Adolescents (13-17 Years Old) With Schizophrenia
Brief Title: Safety and Tolerability of Open-Label Flexible-dose Brexpiprazole as Maintenance Treatment in Adolescents With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 331-10-236
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
Keywords: Brexpiprazole; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- De Novo (Conversion Period) (Experimental): 1-3 milligrams/day (mg/day) brexpiprazole for 1 to 4 weeks
  Interventions: Drug: Brexpiprazole
- Prior and Current Brexpiprazole (Open-label Treatment Period) (Experimental): 1-4 mg/day brexpiprazole; Start at 0.5 mg/day, titrate and maintain between 1mg/day to max of 4 mg/day
  Interventions: Drug: Brexpiprazole
- Prior Aripiprazole and Current Brexpiprazole (Open-label Treatment Period) (Experimental): 1-4 mg/day brexpiprazole; Start at 0.5 mg/day, titrate and maintain between 1mg/day to max of 4 mg/day
  Interventions: Drug: Brexpiprazole
- Prior Placebo and Current Brexpiprazole (Open-label Treatment Period) (Experimental): 1-4 mg/day brexpiprazole; Start at 0.5 mg/day, titrate and maintain between 1mg/day to max of 4 mg/day
  Interventions: Drug: Brexpiprazole
- De Novo (Open-label Treatment Period) (Experimental): 1-4 mg/day brexpiprazole; Start at 0.5 mg/day, titrate and maintain between 1mg/day to max of 4 mg/day
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Once daily, oral tablets
  Other Names: OPC-34712

SUMMARY:
To further characterize the long-term safety and tolerability of brexpiprazole in adolescents with schizophrenia

DETAILED DESCRIPTION:
This is a long-term, multicenter, open-label trial designed to examine the long-term safety and tolerability of brexpiprazole in adolescent participants (ages 13-17) with a DSM-5 diagnosis of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male & female subjects 13-17 years of age, inclusive.
* Subjects who turn 18 during trial 331-10-234 are permitted in this trial.
* Subjects with a current primary diagnosis of schizophrenia, as defined by Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria and confirmed by the K-SADS-PL completed at time of entry into Trial 331-10-234. For de novo subjects who did not participate in Trial 331-10-234, the initial diagnosis of schizophrenia must be made and documented, and the diagnosis confirmed by the K-SADS-PL at screening.
* Subjects who, in the investigator's judgment, require treatment with antipsychotic medication(s).

Exclusion Criteria:

* Subjects with a DSM-5 diagnosis other than schizophrenia that has been the primary focus of treatment within 3 months of screening
* Subjects with a clinical presentation or history that is consistent with delirium, dementia, amnesia, or other cognitive disorders; subjects with psychotic symptoms that are better accounted for by another general medical condition(s) or direct effect of a substance (e.g., medication, illicit drug use).
* History of failure of clozapine treatment or response to clozapine treatment only.
* History of neuroleptic malignant syndrome

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 295 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Guthrie, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (57):
- United States (17):
  - Clinical Research Site #101, Dothan, Alabama
  - Clinical Research Site #128, Anaheim, California
  - Clinical Research Site #105, Culver City, California
  - Clinical Research Site #103, Long Beach, California
  - Clinical Research Site #136, Atlanta, Georgia
  - Clinical Research Site #148, Kansas City, Kansas
  - Clinical Research Site #138, Lake Charles, Louisiana
  - Clinical Research Site #124, Las Vegas, Nevada
  - Clinical Research Site #130, New York, New York
  - Clinical Research Site #100, Rochester, New York
  - Clinical Research Site #121, Kinston, North Carolina
  - Clinical Research Site #133, Cincinnati, Ohio
  - Clinical Research Site #113, Garfield Heights, Ohio
  - Clinical Research Site #102, Oklahoma City, Oklahoma
  - Clinical Research Site #135, Tulsa, Oklahoma
  - Clinical Research Site #140, Frisco, Texas
  - Clinical Research Site #108, Everett, Washington
- Clinical Research Site #321, Nice, France
- Clinical Research Site #283, Naples, Italy
- Mexico (8):
  - Clinical Research Site #163, León, Guanajuato
  - Clinical Research Site #165, Guadalajara, Jalisco
  - Clinical Research Site #171, Monterrey, Nuevo León
  - Clinical Research Site #160, Monterrey, Nuevo León
  - Clinical Research Site #170, San Luis Potosí City, San Luis Potosí
  - Clinical Research Site #161, Culiacán, Sinaloa
  - Clinical Research Site #166, Mérida, Yucatán
  - Clinical Research Site #168, Durango
- Poland (7):
  - Clinical Research Site #263, Tyniec Mały, Dolnyslask
  - Clinical Research Site #266, Bialystok, Podlaskie Voivodeship
  - Clinical Research Site #269, Gdansk, Polorskie
  - Clinical Research Site #260, Poznan
  - Clinical Research Site #272, Poznan
  - Clinical Research Site #270, Wałbrzych
  - Clinical Research Site #267, Wroclaw
- Romania (4):
  - Clinical Research Site #244, Bucharest
  - Clinical Research Site #241, Cluj-Napoca
  - Clinical Research Site #243, Iași
  - Clinical Research Site #242, Timișoara
- Russia (6):
  - Clinical Research Site #542, Arkhangelsk, Primorsky District
  - Clinical Research Site #543, Stavropol, Stavropolskiy Kray
  - Clinical Research Site #545, Moscow
  - Clinical Research Site #541, Saint Petersburg
  - Clinical Research Site #540, Saint Petersburg
  - Clinical Research Site #544, Yaroslavl
- Serbia (5):
  - Clinical Research Site #500, Belgrade
  - Clinical Research Site #504, Belgrade
  - Clinical Research Site #503, Kragujevac
  - Clinical Research Site #502, Niš
  - Clinical Research Site #501, Novi Sad
- Clinical Research Site #224, Torremolinos, Malaga, Spain
- Ukraine (7):
  - Clinical Research Site #526, Poltava, Poltava Oblast
  - Clinical Research Site #527, Dnipro
  - Clinical Research Site #523, Kharkiv
  - Clinical Research Site #521, Kharkiv
  - Clinical Research Site #522, Kherson
  - Clinical Research Site #520, Lviv
  - Clinical Research Site #525, Ternopil

REFERENCES:
- [Derived] Atkinson SD, Shah A, Burgess MV, Hefting N, Chen D, Ward C. Safety and Tolerability of Brexpiprazole in Adolescents With Schizophrenia: A Long-Term, Open-Label Study. JAACAP Open. 2024 May 27;3(2):313-322. doi: 10.1016/j.jaacop.2024.04.005. eCollection 2025 Jun. PMID 40520975

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at multiple sites globally from 23 August 2017 to 22 April 2025. 14 participants underwent a cross-titration and received brexpiprazole for up to 4 weeks in conversion period followed by subsequent enrollment in De-Novo open label treatment (OLT) period.
Pre-assignment Details: Of the 295 participants who were enrolled for the study, 294 participants received the study treatment, and 1 participant did not receive the study drug. All eligible participants who rolled over from the previous study 331-10-234 (NCT03198078), and de novo participants received brexpiprazole tablets during this study.
Groups:
- De Novo (Conversion Period): Participants underwent a cross-titration and received brexpiprazole tablets, orally, once a day (QD), for up to 4 weeks. The dose was increased up to 3 milligrams/day (mg/day) during cross-titration.
- Prior & Current Brexpiprazole (OLT Period): Participants who received brexpiprazole in the previous study 331-10-234, were administered brexpiprazole tablets, orally, once a day (QD) at a starting dose of 0.5 mg/day from Day 1 to Day 4 in this study. Thereafter, the dose was titrated to 1 mg/day by Day 7, with the option of a 1 mg increase or decrease if needed and tolerated. The dose was adjusted within the range of 1 mg/day to 2 mg/day by Day 14, 1 mg/day to 3 mg/day by Day 21, and up to a maximum of 4 mg/day by Day 22 based on clinical judgement. Participants continued to receive flexible dose of brexpiprazole (1 mg/day to 4 mg/day) up to Month 24. Participants were followed for safety for another 21 days. Open-label Treatment Period = OLT Period.
- Prior Aripiprazole & Current Brexpiprazole (OLT Period): Participants who received aripiprazole in the previous study 331-10-234, were administered brexpiprazole tablets, orally, QD at a starting dose of 0.5 mg/day from Day 1 to Day 4 in this study. Thereafter, the dose was titrated to 1 mg/day by Day 7, with the option of a 1 mg increase or decrease if needed and tolerated. The dose was adjusted within the range of 1 mg/day to 2 mg/day by Day 14, 1 mg/day to 3 mg/day by Day 21, and up to a maximum of 4 mg/day by Day 22 based on clinical judgement. Participants continued to receive flexible dose of brexpiprazole (1 mg/day to 4 mg/day) up to Month 24. Participants were followed for safety for another 21 days.
- Prior Placebo & Current Brexpiprazole (OLT Period): Participants who received brexpiprazole or aripiprazole matching placebo tablets in the previous study 331-10-234, were administered brexpiprazole tablets, orally, QD at a starting dose of 0.5 mg/day from Day 1 to Day 4 in this study. Thereafter, the dose was titrated to 1 mg/day by Day 7, with the option of a 1 mg increase or decrease if needed and tolerated. The dose was adjusted within the range of 1 mg/day to 2 mg/day by Day 14, 1 mg/day to 3 mg/day by Day 21, and up to a maximum of 4 mg/day by Day 22 based on clinical judgement. Participants continued to receive flexible dose of brexpiprazole (1 mg/day to 4 mg/day) up to Month 24. Participants were followed for safety for another 21 days.
- De Novo (OLT Period): De novo participants who rolled over from the previous study 331-10-234, and newly enrolled participants in this study were administered brexpiprazole tablets, orally, QD, at a starting dose of 0.5 mg/day from Day 1 to Day 4. Thereafter, the dose was titrated to 1 mg/day by Day 7, with the option of a 1 mg increase or decrease if needed and tolerated. The dose was adjusted within the range of 1 mg/day to 2 mg/day by Day 14, 1 mg/day to 3 mg/day by Day 21, and up to a maximum of 4 mg/day by Day 22 based on clinical judgement. Participants continued to receive flexible dose of brexpiprazole (1 mg/day to 4 mg/day) up to Month 24. Participants were followed for safety for another 21 days.
Period: Conversion Period (4 Weeks)
Arm/Group | De Novo (Conversion Period) | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Started | 14 | 0 | 0 | 0 | 0
Completed | 14 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Open-label Period (About 25 Months)
Arm/Group | De Novo (Conversion Period) | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Started | 0 | 99 | 89 | 87 | 20
Completed | 0 | 58 | 59 | 50 | 11
Not Completed | 0 | 41 | 30 | 37 | 9
Not completed — Adverse Event | 0 | 4 | 2 | 3 | 0
Not completed — Lack of Efficacy | 0 | 4 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 5 | 6 | 3 | 3
Not completed — Non-Compliance With Study Drug | 0 | 1 | 1 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 3 | 0
Not completed — Withdrawal by Participant | 0 | 14 | 8 | 11 | 4
Not completed — Withdrawal by Caregiver | 0 | 10 | 5 | 11 | 1
Not completed — Physician Decision | 0 | 0 | 2 | 0 | 0
Not completed — Reason Not Specified | 0 | 2 | 3 | 4 | 1

BASELINE CHARACTERISTICS:
Population: The enrolled sample consists of all consented/assented participants who were screened for eligibility and deemed eligible.
Groups:
- Prior and Current Brexpiprazole: Participants who received brexpiprazole in the previous study 331-10-234, were administered brexpiprazole tablets, orally, once a day (QD) at a starting dose of 0.5 mg/day from Day 1 to Day 4 in this study. Thereafter, the dose was titrated to 1 mg/day by Day 7, with the option of a 1 mg increase or decrease if needed and tolerated. The dose was adjusted within the range of 1 mg/day to 2 mg/day by Day 14, 1 mg/day to 3 mg/day by Day 21, and up to a maximum of 4 mg/day by Day 22 based on clinical judgement. Participants continued to receive flexible dose of brexpiprazole (1 mg/day to 4 mg/day) up to Month 24. Participants were followed for safety for another 21 days. Open-label Treatment Period = OLT Period.
- Total: Total of all reporting groups
Arm/Group | Prior and Current Brexpiprazole | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period) | Total
Number analyzed (Participants) | 99 | 89 | 87 | 20 | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (1.6) | 15.5 (1.4) | 15.4 (1.5) | 15.5 (1.0) | 15.5 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 49 | 42 | 9 | 153
  Male | 46 | 40 | 45 | 11 | 142
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 65 | 64 | 58 | 18 | 205
  Race: Black or African American | 6 | 2 | 3 | 1 | 12
  Race: American Indian or Alaska Native | 2 | 1 | 4 | 0 | 7
  Race: Asian | 1 | 1 | 0 | 0 | 2
  Race: Native Hawaiin or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Race: Other | 25 | 21 | 21 | 1 | 68
  Race: Missing | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 29 | 25 | 30 | 1 | 85
  Ethnicity: Not Hispanic or Latino | 69 | 64 | 55 | 19 | 207
  Ethnicity: Other | 1 | 0 | 1 | 0 | 2
  Ethnicity: Unknown | 0 | 0 | 0 | 0 | 0
  Ethnicity: Missing | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a clinical trial participant administered a medicinal product and which does not necessarily have a causal relationship with the study treatment.
Time Frame: From the first dose of study drug (including the conversion period and the open-label treatment period in the current study) up to 21 days after the last dose of study drug (up to approximately 25.6 months).
Population: The safety population included all enrolled participants who received at least one dose of the study drug. Participants with conversion were analyzed separately in addition to their analysis in treatment period arms.
Measure: Count of Participants; unit: Participants
Groups:
- Prior & Current Brexpiprazole (OLT Period): Participants who received brexpiprazole in the previous study 331-10-234 were administered brexpiprazole tablets, orally, once a day (QD) at a starting dose of 0.5 mg/day from Day 1 to Day 4 in this study. Thereafter, the dose was titrated to 1 mg/day by Day 7, with the option of a 1 mg increase or decrease if needed and tolerated. The dose was adjusted within the range of 1 mg/day to 2 mg/day by Day 14, 1 mg/day to 3 mg/day by Day 21, and up to a maximum of 4 mg/day by Day 22 based on clinical judgement. Participants continued to receive flexible dose of brexpiprazole (1 mg/day to 4 mg/day) up to Month 24. Participants were followed for safety for another 21 days. Open-label Treatment Period = OLT Period.
Arm/Group | De Novo (Conversion Period) | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 14 | 98 | 89 | 87 | 20
Participants | 5 | 58 | 54 | 63 | 13

2. Primary Outcome: Number of Participants With Serious Treatment Emergent Adverse Events (TEAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical trial participant administered a medicinal product and which does not necessarily have a causal relationship with the study treatment. A serious adverse event (SAE) is any AE occurring at any dose that results in death, life-threatening experience, persistent or significant disability/incapacity, in-patient hospitalization or prolongs hospitalization or congenital anomaly/birth defect. A serious TEAE is defined as an AE that occurred or worsened after the first dose of study treatment up until 30 days after the last dose.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo (Conversion Period) | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 14 | 98 | 89 | 87 | 20
Participants | 0 | 4 | 1 | 3 | 1

3. Primary Outcome: Number of Participants Who Discontinued the Trial Due to AEs
Description: An AE is defined as any untoward medical occurrence in a clinical trial participant administered a medicinal product and which does not necessarily have a causal relationship with the study treatment. Participants who discontinued the trial due to AEs were recorded.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo (Conversion Period) | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 14 | 98 | 89 | 87 | 20
Participants | 0 | 4 | 2 | 3 | 0

4. Secondary Outcome: Mean Change From Baseline in Laboratory Tests (Parameters Assessed in Units Per Liter)
Description: Clinical laboratory assessments included clinical chemistry (alanine aminotransferase [ALT], alkaline phosphatase, aspartate aminotransferase [AST], creatinine phosphokinase (CPK), gamma glutamyl transferase, lactate dehydrogenase.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: The safety population included all enrolled participants who received at least one dose of the study drug. 'Overall number analyzed' indicates the unique participants who were evaluated for this outcome measure. 'Number analyzed' indicates the number of participants evaluable for the specific category. The data for this outcome measure was planned to be collected for only OLT period arm groups.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
units per liter (U/L)
  ALT: number analyzed (Participants) | 91 | 85 | 85 | 20
  ALT | 0.02 (15.35) | 2.09 (10.91) | 0.60 (10.83) | -2.30 (15.13)
  AST: number analyzed (Participants) | 91 | 84 | 85 | 20
  AST | -0.43 (7.20) | 0.12 (8.62) | -0.92 (6.69) | -1.10 (8.35)
  Alkaline Phosphatase: number analyzed (Participants) | 92 | 85 | 85 | 20
  Alkaline Phosphatase | -25.14 (59.48) | -22.36 (60.45) | -13.94 (50.63) | -28.45 (58.93)
  CPK, Total: number analyzed (Participants) | 91 | 85 | 85 | 20
  CPK, Total | -7.12 (114.70) | -17.98 (182.22) | -10.62 (126.12) | -69.70 (283.72)
  Lactate Dehydrogenase: number analyzed (Participants) | 84 | 77 | 83 | 19
  Lactate Dehydrogenase | -1.02 (31.03) | 0.43 (29.70) | -1.75 (26.13) | -6.05 (24.05)
  Gamma Glutamyl Transferase: number analyzed (Participants) | 92 | 85 | 85 | 20
  Gamma Glutamyl Transferase | 0.41 (5.97) | 1.21 (12.73) | 2.22 (13.01) | -0.35 (12.91)

5. Secondary Outcome: Mean Change From Baseline in Laboratory Tests (Parameters Assessed in Milligrams Per Deciliter)
Description: Clinical laboratory assessments included clinical chemistry (bilirubin, urea nitrogen, calcium, glucose, cholesterol including low-density lipoprotein (LDL-C), creatinine, Triglycerides [TG]).
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
milligrams per deciliter (mg/dL)
  Bilirubin: number analyzed (Participants) | 84 | 80 | 78 | 20
  Bilirubin | 0.04 (0.27) | 0.02 (0.25) | -0.05 (0.25) | -0.02 (0.48)
  Calcium: number analyzed (Participants) | 92 | 85 | 85 | 20
  Calcium | -0.07 (0.46) | -0.16 (0.45) | -0.10 (0.34) | 0.00 (0.39)
  Glucose, Fasting: number analyzed (Participants) | 85 | 84 | 81 | 19
  Glucose, Fasting | -0.12 (13.67) | 0.32 (11.32) | 3.11 (16.61) | -2.05 (15.11)
  LDL-C, Fasting: number analyzed (Participants) | 85 | 83 | 79 | 19
  LDL-C, Fasting | 0.46 (27.13) | 7.51 (25.31) | 6.20 (21.44) | 10.11 (30.02)
  Cholesterol, Fasting: number analyzed (Participants) | 87 | 84 | 81 | 19
  Cholesterol, Fasting | 2.68 (32.91) | 8.69 (29.84) | 8.88 (28.02) | 16.89 (35.93)
  TG, Fasting: number analyzed (Participants) | 87 | 84 | 81 | 19
  TG, Fasting | 11.46 (51.00) | 1.32 (57.12) | 2.84 (56.16) | 5.21 (42.45)
  Creatinine: number analyzed (Participants) | 92 | 85 | 85 | 20
  Creatinine | 0.04 (0.14) | 0.02 (0.14) | 0.03 (0.12) | 0.00 (0.12)
  Urea Nitrogen: number analyzed (Participants) | 92 | 85 | 85 | 20
  Urea Nitrogen | 0.50 (3.57) | 0.72 (3.99) | 0.25 (4.85) | 0.60 (4.10)
  Glucose, Urine: number analyzed (Participants) | 94 | 86 | 85 | 20
  Glucose, Urine | -0.01 (0.10) | 0.00 (0.00) | 0.00 (0.08) | 0.00 (0.00)
  Protein, Urine: number analyzed (Participants) | 94 | 86 | 85 | 20
  Protein, Urine | 0.02 (0.49) | -0.13 (0.45) | -0.02 (0.37) | -0.05 (0.32)

6. Secondary Outcome: Mean Change From Baseline in Laboratory Tests (Parameters Assessed in Percentage)
Description: Clinical laboratory assessments of HbA1c are reported in this outcome measure.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage (%) of HbA1c
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
percentage (%) of HbA1c | 0.01 (0.30) | -0.01 (0.32) | 0.05 (0.45) | -0.05 (0.26)

7. Secondary Outcome: Mean Change From Baseline in Laboratory Tests (Parameters Assessed in Million Cells Per Microliter)
Description: Clinical laboratory assessments included hematology including the red blood cell count (RBC Count).
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: million cells/microliter
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
million cells/microliter | 0.09 (0.36) | 0.06 (0.29) | 0.06 (0.33) | 0.01 (0.31)

8. Secondary Outcome: Mean Change From Baseline in Clinical Laboratory Tests (Parameters Assessed in Thousand Cells Per Microliter)
Description: Clinical laboratory assessments included hematology (basophils, eosinophils, neutrophils, leukocytes, lymphocytes, white blood cell (WBC) count, platelets).
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: The safety population included all enrolled participants who received at least one dose of the study drug. Overall number analyzed' indicates the unique participants who were evaluated for this outcome measure. 'Number analyzed' indicates the number of participants evaluable for the specific category. The data for this outcome measure was planned to be collected for only OLT period arm groups.
Measure: Mean (Standard Deviation); unit: thousand cells per microliter
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
thousand cells per microliter
  Basophils: number analyzed (Participants) | 86 | 80 | 80 | 20
  Basophils | 0.00 (0.05) | -0.01 (0.05) | -0.01 (0.05) | 0.01 (0.02)
  Eosinophils: number analyzed (Participants) | 86 | 80 | 80 | 20
  Eosinophils | 0.02 (0.13) | 0.02 (0.11) | -0.01 (0.12) | 0.04 (0.14)
  Lymphocytes: number analyzed (Participants) | 86 | 80 | 80 | 20
  Lymphocytes | 0.07 (0.58) | -0.11 (0.62) | -0.13 (0.58) | 0.02 (0.63)
  Neutrophils: number analyzed (Participants) | 86 | 80 | 80 | 20
  Neutrophils | -0.18 (1.39) | 0.00 (1.48) | -0.05 (1.79) | -0.44 (1.32)
  WBC: number analyzed (Participants) | 86 | 80 | 80 | 20
  WBC | -0.08 (1.53) | -0.09 (1.87) | -0.22 (1.99) | -0.35 (1.35)
  Platelets: number analyzed (Participants) | 85 | 80 | 80 | 20
  Platelets | -2.67 (59.28) | -11.01 (43.48) | -5.05 (56.07) | 19.20 (55.50)

9. Secondary Outcome: Mean Change From Baseline in Laboratory Tests (Parameters That Were Unitless)
Description: Clinical laboratory assessments of pH are reported in this outcome measure.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
unitless | 0.04 (0.63) | -0.06 (0.51) | 0.03 (0.60) | 0.05 (0.69)

10. Secondary Outcome: Mean Change From Baseline in Laboratory Tests (Parameters Assessed in Nanograms Per Milliliter)
Description: Clinical laboratory assessments included prolactin for both males and females.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/ml)
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 93 | 85 | 85 | 19
nanograms per milliliter (ng/ml)
  Prolactin - Females: number analyzed (Participants) | 50 | 47 | 41 | 8
  Prolactin - Females | -8.34 (15.27) | 9.86 (10.24) | 6.07 (21.14) | -1.73 (9.41)
  Prolactin - Males: number analyzed (Participants) | 43 | 38 | 44 | 11
  Prolactin - Males | 0.83 (12.56) | 7.70 (8.82) | 2.42 (12.86) | -0.79 (23.91)

11. Secondary Outcome: Mean Change From Baseline in Laboratory Tests (Parameters Assessed in Milliequivalents Per Liter)
Description: Clinical laboratory assessments including chloride and potassium are reported in this outcome measure.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milliequivalents per liter (mEq/dL)
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
milliequivalents per liter (mEq/dL)
  Chloride: number analyzed (Participants) | 92 | 85 | 85 | 20
  Chloride | 0.16 (2.56) | -0.35 (2.77) | 0.19 (3.18) | 0.45 (3.59)
  Potassium: number analyzed (Participants) | 92 | 85 | 85 | 20
  Potassium | 0.02 (0.36) | -0.09 (0.46) | 0.02 (0.45) | 0.04 (0.37)

12. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Tests
Description: Laboratory assessments included hematology, chemistry, and urinalysis. Abnormality criteria included: In mg/dL [high bilirubin≥2.0, low calcium≤8.2, high cholesterol fasting≥240, HDL-C, Fasting<40 male(M)/ < 50 female(F); LDL-C, fasting≥160, high glucose, fasting≥100, non-fasting≥200 high TG, fasting≥150, high urate≥8.5 F/≥10.5 M, high protein urine≥2 units increase]; high creatine kinase(units per liter [U/L])>3xupper limit of normal (ULN)]; high eosinophils/leukocytes ≥10%;ALT>3×ULN; in mEq/L [Cl≤ 90; potassium≤ 2.5; sodium low≤ 126, high ≥156]; platelets≤75000/mm3; hemoglobin≤11g/dL M/≤ 9.5 F; glucose, urine≥2 units inc.; casts≥2 units inc.; hematocrit≤37% and decrease of≥3% points, M/≤ 32% and ≥3% points dec.,F. Number of participants with clinically significant laboratory test abnormalities were reported as per criteria defined in protocol. The categories with at least 1 participant with clinically significant abnormalities are reported.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
Participants
  ALT: High: number analyzed (Participants) | 95 | 87 | 85 | 20
  ALT: High | 1 | 1 | 0 | 1
  Bilirubin: High: number analyzed (Participants) | 92 | 86 | 85 | 20
  Bilirubin: High | 2 | 0 | 0 | 0
  Calcium: Low: number analyzed (Participants) | 95 | 87 | 85 | 20
  Calcium: Low | 1 | 3 | 0 | 0
  Chloride: Low: number analyzed (Participants) | 95 | 87 | 85 | 20
  Chloride: Low | 1 | 0 | 1 | 0
  Cholesterol, Fasting: High: number analyzed (Participants) | 94 | 87 | 83 | 19
  Cholesterol, Fasting: High | 2 | 1 | 5 | 3
  Creatine Kinase: High: number analyzed (Participants) | 95 | 87 | 85 | 20
  Creatine Kinase: High | 8 | 9 | 4 | 0
  Glucose, Fasting: High: number analyzed (Participants) | 94 | 87 | 83 | 19
  Glucose, Fasting: High | 29 | 26 | 18 | 9
  HDL Cholesterol, Fasting: Low: number analyzed (Participants) | 94 | 87 | 83 | 19
  HDL Cholesterol, Fasting: Low | 25 | 21 | 17 | 2
  LDL-C, Fasting: High: number analyzed (Participants) | 94 | 87 | 83 | 19
  LDL-C, Fasting: High | 3 | 0 | 3 | 2
  Potassium: Low: number analyzed (Participants) | 95 | 87 | 85 | 20
  Potassium: Low | 1 | 0 | 0 | 0
  Sodium: Low: number analyzed (Participants) | 95 | 87 | 85 | 20
  Sodium: Low | 0 | 0 | 1 | 0
  Sodium: High: number analyzed (Participants) | 95 | 87 | 85 | 20
  Sodium: High | 1 | 0 | 0 | 0
  TG,Fasting: High: number analyzed (Participants) | 94 | 87 | 83 | 19
  TG,Fasting: High | 21 | 23 | 20 | 5
  Urate: High: number analyzed (Participants) | 95 | 87 | 85 | 20
  Urate: High | 1 | 0 | 0 | 0
  Eosinophils/Leukocytes: High: number analyzed (Participants) | 94 | 86 | 85 | 20
  Eosinophils/Leukocytes: High | 0 | 2 | 1 | 0
  Hematocrit: Low: number analyzed (Participants) | 91 | 86 | 84 | 20
  Hematocrit: Low | 2 | 3 | 2 | 0
  Hemoglobin: Low: number analyzed (Participants) | 94 | 86 | 85 | 20
  Hemoglobin: Low | 1 | 4 | 3 | 0
  Platelets: Low: number analyzed (Participants) | 94 | 86 | 85 | 20
  Platelets: Low | 1 | 0 | 0 | 0
  Glucose, Urine: High: number analyzed (Participants) | 95 | 87 | 85 | 20
  Glucose, Urine: High | 2 | 0 | 1 | 0
  Protein, Urine: High: number analyzed (Participants) | 95 | 87 | 85 | 20
  Protein, Urine: High | 1 | 0 | 1 | 0
  Prolactin: High: number analyzed (Participants) | 95 | 87 | 85 | 20
  Prolactin: High | 23 | 29 | 27 | 8

13. Secondary Outcome: Mean Change From Baseline in Vital Signs (Parameters Assessed in Beats Per Minute)
Description: Vital sign measurements included pulse rate assessed in beats per minute in standing and supine position.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: The safety population included all enrolled participants who received at least one dose of the study drug. The data for this outcome measure was planned to be collected for only OLT period arm groups.
Measure: Mean (Standard Deviation); unit: beats per minute (beats/min)
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
beats per minute (beats/min)
  Pulse Rate: Standing | -0.6 (12.8) | -1.9 (10.0) | -0.5 (10.6) | -2.8 (11.0)
  Pulse Rate: Supine | 1.1 (10.2) | -1.6 (10.1) | -0.5 (14.5) | 0.7 (11.7)

14. Secondary Outcome: Mean Change From Baseline in Vital Signs (Parameters Assessed in Millimeters of Mercury)
Description: Vital sign measurements included systolic blood pressure (SBP) and diastolic blood pressure (DBP). Blood pressure measurements were made in the supine and standing positions after the participant has been in each position at least 3 minutes.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: The safety population included all enrolled participants who received at least one dose of the study drug. 'Overall number analyzed' indicates the unique participants who were evaluated for this outcome measure. The data for this outcome measure was planned to be collected for only OLT period arm groups.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
millimeters of mercury (mmHg)
  SBP: Standing | 0.7 (9.0) | 0.5 (9.6) | 1.5 (10.8) | -1.7 (6.5)
  SBP: Supine | 0.7 (8.9) | 0.4 (9.5) | 2.1 (11.5) | -0.3 (6.8)
  DBP: Standing | 0.2 (7.7) | 1.2 (8.5) | 0.2 (8.3) | 0.1 (6.7)
  DBP: Supine | 0.8 (8.5) | 0.4 (7.4) | -0.5 (7.5) | 0.4 (8.9)

15. Secondary Outcome: Mean Change From Baseline in Vital Signs (Parameters Assessed in Centimeters)
Description: Vital sign measurements included height assessed in centimeters.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
centimeters (cm) | 1.4 (5.4) | 2.4 (4.5) | 2.0 (4.2) | 3.5 (4.2)

16. Secondary Outcome: Mean Change From Baseline in Vital Signs (Parameters Assessed in Kilograms)
Description: Vital sign measurements included weight assessed in kilograms.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
kilograms (kg) | 3.8 (5.8) | 4.2 (7.5) | 3.8 (6.6) | 3.4 (4.3)

17. Secondary Outcome: Mean Change From Baseline in Vital Signs (Parameters Assessed in Celsius)
Description: Vital sign measurements included temperature assessed in celsius.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: celsius (°C)
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
celsius (°C) | -0.0 (0.4) | -0.0 (0.3) | -0.0 (0.4) | 0.0 (0.3)

18. Secondary Outcome: Mean Change From Baseline in Vital Signs (Parameters Assessed in Z-Score)
Description: Vital sign measurements- Z-score for body weight (BW), height, and BMI. To adjust for normal growth, z-scores were derived, which normalize for the natural growth of pediatric patients and adolescents. Z-score was calculated as the deviation of the participant's each parameter from the mean for the respective parameter of the reference population divided by the standard deviation (SD) for the reference population. Z-score-0 represents the population mean for the respective parameter. Positive Z-scores-values above the mean, negative Z-scores indicate values below the mean. BW and BMI: Higher Z-scores-Potential overweight/obesity (worse outcome if excessive). Lower Z-scores -Underweight (worse outcome if extreme). Height: Higher Z-scores-Taller than average (neutral unless clinically relevant). Lower Z-scores → Short stature (may indicate growth issues). Z ≥ +2-Above normal range (e.g., overweight or obesity for BMI). Z ≤ -2-Below normal range (e.g., underweight or short stature).
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
z-score
  Z-Score of Body Weight | -0.0 (0.5) | -0.0 (0.5) | 0.0 (0.5) | 0.0 (0.4)
  Z-Score of Height: number analyzed (Participants) | 93 | 80 | 84 | 20
  Z-Score of Height | -0.1 (0.8) | 0.1 (0.5) | 0.0 (0.5) | 0.3 (0.6)
  Z-Score of BMI: number analyzed (Participants) | 93 | 80 | 84 | 20
  Z-Score of BMI | 0.0 (0.6) | -0.1 (0.6) | 0.0 (0.6) | -0.1 (0.5)

19. Secondary Outcome: Mean Change From Baseline in Vital Signs (Parameters Assessed in Kilograms Per Meter Square)
Description: Vital sign measurements included body mass index (BMI).
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
kilograms per meter square (kg/m^2) | 1.0 (2.3) | 0.9 (2.8) | 0.8 (2.2) | 0.1 (2.2)

20. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital sign measurements included SBP, and DBP, pulse rate, body temperature, body weight, BMI, and height. Vital sign measurements included pulse rate in supine and standing positions (low: <50 beats per minute [bpm] and decrease ≥15 bpm; High: >120 bpm and increase ≥15 bpm), SBP in supine and standing positions (low: <110 mmHg and decrease ≥20 mmHg; High: >120 mmHg and increase ≥20 mmHg), DBP in supine and standing positions (low: <60 mmHg and decrease ≥15 mmHg; High: >80 mmHg and increase ≥15 mmHg), weight in kg (low: ≥7% decrease; High: ≥7% increase), orthostatic hypotension, (≥20mmHg decrease in SBP or ≥10 mmHg in DBP in heart rate from supine to standing). Number of participants with clinically significant abnormalities in vital signs were reported as per criteria defined in protocol. The categories with at least one participant with clinically significant abnormalities in vital signs are reported.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
Participants
  SBP, Standing: Low | 7 | 5 | 6 | 0
  SBP, Standing: High | 10 | 11 | 14 | 2
  SBP, Supine: Low | 9 | 7 | 5 | 0
  SBP, Supine: High | 3 | 8 | 9 | 0
  DBP, Standing: Low | 1 | 5 | 1 | 1
  DBP, Standing: High | 14 | 14 | 18 | 3
  DBP, Supine: Low | 6 | 3 | 3 | 2
  DBP, Supine: High | 12 | 11 | 8 | 0
  Pulse Rate, Standing: High | 0 | 0 | 1 | 0
  Pulse Rate, Supine: Low | 0 | 0 | 1 | 0
  Pulse Rate, Supine: High | 0 | 0 | 1 | 0
  Weight: Low | 9 | 5 | 9 | 1
  Weight: High | 46 | 40 | 40 | 13
  Orthostatic Hypotension: Low | 16 | 23 | 12 | 2

21. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) (Parameters Assessed in Milliseconds)
Description: 12-lead ECG recordings were obtained for parameters including PR interval, QRS duration, QT interval, QTcB [QT interval as corrected for heart rate by Bazett's formula] interval, QTcF [QT interval as corrected for heart rate by Fridericia's formula] interval, QTcN [QT interval corrected for heart rate by the FDA Neuropharm] interval, and RR interval.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
milliseconds (ms)
  PR Interval: number analyzed (Participants) | 96 | 86 | 84 | 20
  PR Interval | 4.2 (14.4) | 2.5 (14.3) | 3.6 (15.6) | -2.0 (16.2)
  QRS Duration: number analyzed (Participants) | 96 | 86 | 84 | 20
  QRS Duration | 1.6 (8.1) | 1.5 (7.8) | 0.8 (6.8) | 1.1 (10.1)
  QT Interval: number analyzed (Participants) | 96 | 86 | 84 | 20
  QT Interval | 4.8 (27.9) | 5.6 (28.0) | 1.3 (26.7) | 1.6 (27.8)
  QTCB Interval: number analyzed (Participants) | 96 | 86 | 84 | 20
  QTCB Interval | -0.9 (26.5) | -0.1 (25.2) | -0.8 (28.6) | 5.6 (20.5)
  QTCF Interval: number analyzed (Participants) | 96 | 86 | 84 | 20
  QTCF Interval | 1.1 (19.6) | 1.8 (20.8) | -0.1 (21.9) | 4.1 (16.4)
  QTCN Interval: number analyzed (Participants) | 96 | 86 | 84 | 20
  QTCN Interval | 0.7 (20.4) | 1.5 (21.2) | -0.3 (22.9) | 4.3 (16.6)
  RR Interval: number analyzed (Participants) | 96 | 86 | 84 | 20
  RR Interval | 26.9 (175.1) | 26.5 (146.1) | 10.0 (166.0) | -12.3 (147.7)

22. Secondary Outcome: Mean Change From Baseline in ECG Parameters (Parameters Assessed in Beats Per Minute)
Description: Twelve-lead ECG recordings were obtained for parameters including mean heart rate.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
beats/min | -2.1 (14.7) | -1.7 (13.3) | -0.8 (13.8) | 1.8 (13.6)

23. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in ECG Parameters
Description: 12-lead ECG recordings were obtained for certain parameters and the 12-lead ECG abnormality criteria included bradycardia ≤ 50 bpm and decrease ≥15 bpm; sinus bradycardia ≤ 50 bpm and decrease of ≥ 15 bpm, supraventricular premature beat (SVPB)-not present at baseline and present post baseline, ventricular premature beat (VPB)- not present at baseline and present post baseline; and primary (1°) atrioventricular (AV) block (PR ≥200 milliseconds [msec] and increase of ≥50 msec, right bundle-branch block (RBBB) and symmetrical T-wave inversion (Sym T Wave Inv) - both not present at baseline and present post baseline; Increase in QTc-QTcF ≥ 450 msec for males, ≥ 470 msec for females. Number of participants with clinically significant ECG abnormalities was reported as per the criteria defined in the protocol. The categories with at least 1 participant with clinically significant ECG abnormalities are reported.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
Participants
  Bradycardia: number analyzed (Participants) | 96 | 86 | 84 | 20
  Bradycardia | 4 | 1 | 1 | 0
  Sinus Bradycardia: number analyzed (Participants) | 96 | 86 | 84 | 20
  Sinus Bradycardia | 4 | 1 | 1 | 0
  SVPB: number analyzed (Participants) | 96 | 86 | 84 | 20
  SVPB | 1 | 1 | 2 | 0
  VPB: number analyzed (Participants) | 95 | 87 | 85 | 20
  VPB | 1 | 1 | 0 | 0
  1° AV Block: number analyzed (Participants) | 96 | 86 | 84 | 20
  1° AV Block | 1 | 2 | 0 | 0
  RBBB: number analyzed (Participants) | 96 | 87 | 85 | 20
  RBBB | 1 | 0 | 1 | 0
  Sym T-Wave Inv: number analyzed (Participants) | 96 | 87 | 85 | 20
  Sym T-Wave Inv | 0 | 0 | 0 | 1
  QT: number analyzed (Participants) | 96 | 86 | 84 | 20
  QT | 1 | 0 | 0 | 0
  Increase in QTcF: number analyzed (Participants) | 96 | 86 | 84 | 20
  Increase in QTcF | 0 | 1 | 0 | 0

24. Secondary Outcome: Mean Change From Baseline on the Abnormal Involuntary Movement Scale (AIMS) Total Score
Description: The AIMS assessment consists of 12 items rating the involuntary movements: Facial and oral movements (4 items), extremity movements (2 items), and trunk movements (1 item) were observed unobtrusively while the participant is at rest and the investigator also made global judgments on the participant's dyskinesias (2 items), and dental status (2 items). Severity of each item was rated on a 5-point scale, with a score of 0 (absence of symptoms) to 4 (severe condition). Total Score is the sum of the scores of all 12 items, ranging from 0 to 48, higher scores indicate severe condition. A negative change reflects an improvement or reduction in the severity of abnormal movements.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
score on a scale | -0.01 (0.30) | -0.06 (0.35) | 0.09 (0.68) | -0.05 (0.22)

25. Secondary Outcome: Mean Change From Baseline on the Simpson-Angus Scale (SAS) Total Score
Description: The SAS consists of a list of 10 symptoms of Parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia). Each item is rated on a 5-point scale, with a score of zero representing absence of symptoms, and a score of 4 representing a severe condition. The SAS Total Score is the sum of the scores for all 10 items, ranging from 0-40. A negative change reflects an improvement or reduction in Parkinsonism severity.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
score on a scale | -0.18 (0.69) | -0.33 (0.77) | 0.17 (1.40) | -0.75 (2.38)

26. Secondary Outcome: Mean Change From Baseline in the Barnes Akathisia Rating Scale (BARS) Total Score
Description: The BARS score is based only on the item of "Global Clinical Assessment of Akathisia". The BARS consists of 4 items related to akathisia as follows. Item 1: objective observation of akathisia by the investigator; Item 2: subjective feelings of restlessness by the participant; Item 3: subjective distress due to akathisia; and Item 4: global clinical assessment of akathisia. The first 3 items will be rated on a 4-point Likert scale from 0 to 3, with 0 representing absence of symptoms and 3 representing a severe condition. The BARS global clinical assessment score refers to the ratings from the 4th item Global Clinical Assessment of Akathisia, which is a 6-point Likert scale from 0 to 5, with 0 representing absence of symptoms and 5 representing severe akathisia. Total score is the sum of the scores of all 4 items, ranging from 0 to 14. Higher score indicates severe akathisia. A negative change from baseline reflects improvement or reduction in the severity of akathisia symptoms.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
score on a scale | -0.02 (0.29) | -0.08 (0.34) | 0.02 (0.53) | -0.15 (0.49)

27. Secondary Outcome: Number of Participants With At Least One Occurrence of Suicidal Behavior or Suicidal Ideation as Recorded on Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a scale used to report at least one occurrence of any suicidal behavior or suicidal ideation. Suicidal behavior was defined as reporting any of the following items: actual attempt, interrupted attempt, aborted attempt, and preparatory acts or behavior. The suicidal ideation total score is the sum of intensity scores of 5 items (frequency, duration, controllability, deterrents, and reasons for ideation). The score of each intensity item ranges from 0 (none) to 5 (worst) and the total score ranges from 0 to 25. Lower scores indicate improvement.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo (Conversion Period) | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 14 | 98 | 89 | 87 | 20
Participants | 0 | 5 | 4 | 6 | 1

28. Secondary Outcome: Number of Participants With Psychotropic Side Effects as Assessed by Udvalg for Kliniske Undersogelser (UKU) Rating Scale
Description: The UKU rating scale is a semi-structured interview used to assess the side effects of participants being treated with antipsychotic drugs. Each item (i.e., each symptom) of the UKU side effects is defined by the means of a 4-point-scale (0-1-2-3) if it is assessed in psychic, autonomic (auto), neurologic, other categories. In general, Degree 0 means "doubtfully or not present (NP)", and Degrees 1, 2, and 3 indicate that the symptom is present to a mild, moderate or severe degree, respectively.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
Participants
  Psychic: Concentration Difficulties: NP | 38 | 30 | 32 | 2
  Psychic: Concentration Difficulties: Mild | 30 | 30 | 33 | 9
  Psychic: Concentration Difficulties: Moderate | 29 | 24 | 20 | 8
  Psychic: Concentration Difficulties: Severe | 1 | 5 | 2 | 1
  Psychic: Asthenia/Lassitude: NP | 59 | 49 | 44 | 5
  Psychic: Asthenia/Lassitude: Mild | 26 | 24 | 30 | 9
  Psychic: Asthenia/Lassitude: Moderate | 13 | 16 | 13 | 6
  Psychic: Sleepiness/Sedation: NP | 77 | 65 | 63 | 9
  Psychic: Sleepiness/Sedation: Mild | 16 | 20 | 23 | 10
  Psychic: Sleepiness/Sedation: Moderate | 5 | 4 | 1 | 1
  Psychic: Failing Memory, Degree: NP | 56 | 51 | 49 | 9
  Psychic: Failing Memory: Mild | 28 | 21 | 27 | 5
  Psychic: Failing Memory: Moderate | 14 | 17 | 11 | 6
  Psychic: Depression: NP | 60 | 49 | 46 | 7
  Psychic: Depression: Mild | 31 | 26 | 31 | 7
  Psychic: Depression: Moderate | 6 | 13 | 10 | 6
  Psychic: Depression: Severe | 1 | 1 | 0 | 0
  Psychic: Tension/Lnner Unrest: NP | 46 | 37 | 35 | 5
  Psychic: Tension/Lnner Unrest: Mild | 36 | 32 | 35 | 13
  Psychic: Tension/Lnner Unrest: Moderate | 15 | 20 | 15 | 1
  Psychic: Tension/Lnner Unrest: Severe | 1 | 0 | 2 | 1
  Psychic: Increased Duration Of Sleep: NP | 82 | 79 | 73 | 13
  Psychic: Increased Duration Of Sleep: Mild | 16 | 7 | 12 | 6
  Psychic: Increased Duration Of Sleep: Moderate | 0 | 3 | 2 | 1
  Psychic: Reduced Duration Of Sleep, Degree: NP | 88 | 69 | 68 | 12
  Psychic: Reduced Duration Of Sleep: Mild | 7 | 15 | 18 | 5
  Psychic: Reduced Duration Of Sleep: Moderate | 2 | 5 | 1 | 3
  Psychic: Reduced Duration Of Sleep: Severe | 1 | 0 | 0 | 0
  Psychic: Inc. Dream Activity: NP | 88 | 75 | 74 | 15
  Psychic: Inc. Dream Activity: Mild | 10 | 11 | 11 | 5
  Psychic: Inc. Dream Activity: Moderate | 0 | 3 | 2 | 0
  Psychic: Emotional Indifference: NP | 45 | 47 | 48 | 3
  Psychic: Emotional Indifference: Mild | 33 | 24 | 22 | 7
  Psychic: Emotional Indifference: Moderate | 20 | 17 | 15 | 10
  Psychic: Emotional Indifference: Severe | 0 | 1 | 2 | 0
  Neurologic: Dystonia: NP | 94 | 88 | 85 | 20
  Neurologic: Dystonia: Mild | 3 | 1 | 2 | 0
  Neurologic: Dystonia: Moderate | 1 | 0 | 0 | 0
  Neurologic: Rigidity: Not Present | 94 | 87 | 81 | 17
  Neurologic: Rigidity: Mild | 4 | 2 | 6 | 3
  Neurologic: Hypokinesia/Akinesia: NP | 93 | 85 | 82 | 19
  Neurologic: Hypokinesia/Akinesia: Mild | 5 | 4 | 4 | 1
  Neurologic: Hypokinesia/Akinesia: Moderate | 0 | 0 | 1 | 0
  Neurologic: Hyperkinesia Logic: NP | 96 | 89 | 85 | 20
  Neurologic: Hyperkinesia Logic: Mild | 1 | 0 | 2 | 0
  Neurologic: Hyperkinesia Logic: Moderate | 1 | 0 | 0 | 0
  Neurologic: Tremor: Not Present | 86 | 83 | 75 | 17
  Neurologic: Tremor: Mild | 11 | 5 | 10 | 3
  Neurologic: Tremor: Moderate | 1 | 1 | 2 | 0
  Neurologic: Akathisia: Not Present | 93 | 77 | 74 | 19
  Neurologic: Akathisia: Mild | 4 | 9 | 11 | 1
  Neurologic: Akathisia: Moderate | 1 | 3 | 2 | 0
  Neurologic: Epileptic Seizures: NP | 98 | 89 | 87 | 20
  Neurologic: Paraesthesias: NP | 98 | 87 | 85 | 20
  Neurologic: Paraesthesias: Mild | 0 | 2 | 2 | 0
  Auto:Accommodation Disturbances :NP | 98 | 87 | 85 | 16
  Auto: Accommodation Disturbances: Mild | 0 | 1 | 2 | 0
  Auto: Accommodation Disturbances: Moderate | 0 | 1 | 0 | 4
  Auto: Increased Salivation: Not Present | 95 | 84 | 81 | 20
  Auto: Increased Salivation: Mild | 3 | 4 | 3 | 0
  Auto: Increased Salivation: Moderate | 0 | 0 | 3 | 0
  Auto: Increased Salivation: Severe | 0 | 1 | 0 | 0
  Auto: Reduced Salivation: Not Present | 98 | 88 | 83 | 19
  Auto: Reduced Salivation: Mild | 0 | 1 | 4 | 1
  Auto: Nausea/Vomiting: Not Present | 93 | 86 | 76 | 19
  Auto: Nausea/Vomiting: Mild | 4 | 2 | 9 | 1
  Auto: Nausea/Vomiting: Moderate | 1 | 1 | 1 | 0
  Auto: Nausea/Vomiting: Severe | 0 | 0 | 1 | 0
  Auto: Diarrhoea: Not Present | 97 | 88 | 84 | 20
  Auto: Diarrhoea: Mild | 1 | 0 | 2 | 0
  Auto: Diarrhoea: Moderate | 0 | 1 | 1 | 0
  Auto: Constipation: Not Present | 95 | 87 | 85 | 17
  Auto: Constipation: Mild | 2 | 2 | 2 | 3
  Auto: Constipation: Moderate | 1 | 0 | 0 | 0
  Auto: Micturition Disturbances: NP | 97 | 88 | 85 | 20
  Auto: Micturition Disturbances: Mild | 1 | 1 | 1 | 0
  Auto: Micturition Disturbances: Moderate | 0 | 0 | 1 | 0
  Auto: Polyuria/Polydipsia: Not Present | 97 | 85 | 84 | 20
  Auto:Polyuria/Polydipsia, Degree:Mild | 0 | 4 | 1 | 0
  Auto:Polyuria/Polydipsia:Moderate | 1 | 0 | 2 | 0
  Auto:Orthostatic Dizziness: Not Present | 95 | 84 | 81 | 17
  Auto:Orthostatic Dizziness: Mild | 3 | 5 | 5 | 3
  Auto:Orthostatic Dizziness: Moderate | 0 | 0 | 1 | 0
  Auto:Palpitations/Tachycardia:Not Present | 94 | 85 | 82 | 17
  Auto:Palpitations/Tachycardia:Mild | 3 | 4 | 3 | 3
  Auto:Palpitations/Tachycardia:Moderate | 1 | 0 | 1 | 0
  Auto:Palpitations/Tachycardia:Severe | 0 | 0 | 1 | 0
  Auto:Inc. Tendency To Sweat:NP | 84 | 19 | 84 | 19
  Auto:Inc. Tendency To Sweat:Mild | 2 | 1 | 3 | 1
  Auto:Inc. Tendency To Sweat:Moderate | 0 | 0 | 0 | 0
  Auto:Inc. Tendency To Sweat:Severe | 1 | 0 | 1 | 0
  Other:Rash:Not Present | 98 | 89 | 87 | 20
  Other:Morbilliform: Mild | 2 | 0 | 0 | 0
  Other:Petechial: Mild | 2 | 0 | 0 | 0
  Other: Urticarial: Mild | 2 | 0 | 1 | 0
  Other:Psoriatic: Mild | 2 | 0 | 0 | 0
  Other:Cannot Be Classified: Mild | 2 | 0 | 1 | 1
  Other:Pruritus, Degree: Not Present | 98 | 87 | 85 | 20
  Other:Pruritus: Mild | 0 | 1 | 1 | 0
  Other:Pruritus: Moderate | 0 | 1 | 1 | 0
  Other:Photosensitivity: Not Present | 97 | 86 | 86 | 20
  Other:Photosensitivity : Mild | 1 | 3 | 1 | 0
  Other:Inc. Pigmentation: NP | 98 | 89 | 87 | 20
  Other:Weight Gain: Not Present | 74 | 66 | 67 | 11
  Other:Weight Gain: Mild | 16 | 15 | 15 | 6
  Other:Weight Gain: Moderate | 18 | 6 | 5 | 3
  Other:Weight Gain: Severe | 0 | 2 | 0 | 0
  Other:Weight Loss: Not Present | 80 | 77 | 76 | 15
  Other:Weight Loss: Mild | 15 | 11 | 9 | 5
  Other:Weight Loss: Moderate | 3 | 1 | 2 | 0
  Other: Menorrhagia: NP: number analyzed (Participants) | 70 | 65 | 63 | 16
  Other: Menorrhagia: NP | 70 | 64 | 61 | 16
  Other:Menorrhagia:Mild: number analyzed (Participants) | 70 | 65 | 63 | 16
  Other:Menorrhagia:Mild | 0 | 1 | 1 | 0
  Other:Menorrhagia:Severe: number analyzed (Participants) | 70 | 64 | 63 | 16
  Other:Menorrhagia:Severe | 0 | 0 | 1 | 0
  Other: Amenorrhoea: NP: number analyzed (Participants) | 69 | 61 | 58 | 14
  Other: Amenorrhoea: NP | 68 | 58 | 57 | 14
  Other:Amenorrhoea:Mild: number analyzed (Participants) | 69 | 61 | 58 | 14
  Other:Amenorrhoea:Mild | 1 | 1 | 1 | 0
  Other:Amenorrhoea: Moderate: number analyzed (Participants) | 69 | 61 | 58 | 14
  Other:Amenorrhoea: Moderate | 0 | 1 | 0 | 0
  Other:Amenorrhoea:Severe: number analyzed (Participants) | 69 | 61 | 58 | 14
  Other:Amenorrhoea:Severe | 0 | 1 | 0 | 0
  Other:Galactorrhoea : Not Present | 88 | 78 | 75 | 20
  Other:Galactorrhoea : Mild | 0 | 1 | 0 | 0
  Other: Gynaecomastia: NP | 77 | 70 | 70 | 17
  Other: Inc. Sexual Desire: Not Present | 91 | 84 | 83 | 19
  Other: Inc. Sexual Desire: Mild | 0 | 1 | 2 | 1
  Other: Inc. Sexual Desire: Moderate | 1 | 0 | 0 | 0
  Other:Diminished Sexual Desire: NP | 91 | 80 | 81 | 14
  Other:Diminished Sexual Desire: Mild | 1 | 5 | 2 | 5
  Other:Diminished Sexual Desire: Moderate | 0 | 0 | 2 | 0
  Other:Diminished Sexual Desire: Severe | 0 | 0 | 0 | 1
  Other:Erectile Dysfunction: NP | 66 | 53 | 63 | 10
  Other:Erectile Dysfunction: Mild | 0 | 3 | 0 | 2
  Other:Ejaculatory Dysfunction:Not Present | 65 | 54 | 62 | 12
  Other:Ejaculatory Dysfunction:Mild | 0 | 1 | 0 | 0
  Other:Ejaculatory Dysfunction:Moderate | 0 | 1 | 0 | 0
  Other:Orgastic Dysfunction: NP | 88 | 83 | 82 | 19
  Other:Orgastic Dysfunction: Mild | 0 | 1 | 1 | 1
  Other : Dry Vagina, Degree : Not Present | 67 | 66 | 62 | 14
  Other: Headache : Not Present | 98 | 89 | 87 | 20
  Other:Tension Headache: Mild | 2 | 4 | 5 | 3
  Other:Tension Headache: Moderate | 2 | 0 | 0 | 1
  Other:Migraine: Mild | 3 | 2 | 5 | 0
  Other:Other Forms: Mild | 3 | 1 | 5 | 0
  Other:Other Forms: Moderate | 0 | 1 | 83 | 13
  Other:Physical Dependence:NP | 93 | 83 | 83 | 13
  Other:Physical Dependence:Mild | 0 | 0 | 0 | 1
  Other:Physical Dependence:Moderate | 0 | 0 | 0 | 2
  Other:Psychic Dependence: NP | 98 | 88 | 86 | 17
  Other:Psychic Dependence:Mild | 0 | 0 | 1 | 1
  Other:Psychic Dependence:Moderate | 0 | 0 | 0 | 2

29. Secondary Outcome: Number of Participants With at Least One Occurrence of Cognitive Adverse Effects Assessed by New York Assessment for Adverse Cognitive Effects of Neuropsychiatric Treatment (NY-AACENT)
Description: The NY-AACENT is used to detect changes in cognitive function for neurological or psychiatric problems, specifically created to be used in pediatric population (ages 12 -17), but could be used with other age groups, as appropriate. Each of the 7 items is derived from the 7 domains as follows: Working Memory, Attention/Vigilance, Verbal Learning/Memory, Visual Learning/Memory, Reasoning and Problem Solving, Speed of Processing, and Social Cognition. Each score is derived as follows: 0=not present in the past week; 1=present (during past week) and mild; 2=present (during past week) and moderate; 3=present (during past week) and severe; and 4=present (during past week) and extreme; and the item score is set to missing/unknown. The NY-AACENT total score is calculated by summing up 7 individual item scores at participant-visit level. The Total range is 0-28. Higher scores reflects greater severity and frequency of cognitive problems and lower scores shows absence or mild cognitive issues.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
Participants
  Working Memory | 69 | 57 | 61 | 14
  Attention/Vigilance | 77 | 72 | 69 | 17
  Verbal Learning | 59 | 46 | 51 | 17
  Visual Learning | 35 | 33 | 35 | 5
  Reasoning | 76 | 69 | 65 | 18
  Speed of Processing | 72 | 59 | 59 | 15
  Social Cognition | 77 | 71 | 64 | 17
  Any Sign/Symptoms | 88 | 78 | 74 | 20

30. Secondary Outcome: Number of Participants With Stages of Tanner Scale Score at Baseline and Month 24
Description: The Tanner scale is a classification system used to assess physical development during puberty, detailing five distinct stages of growth. The Tanner Staging Scale assessment consists of 2 domains for girls and 3 domains for boys. Participants with change in Tanner Staging Scale (Stage 1-5) Score are reported.
Time Frame: Baseline, Month 24
Population: The safety population included all enrolled participants who received at least one dose of the study drug. Number analyzed are the participants with data available at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 98 | 89 | 87 | 20
Participants
  Boys: Baseline-Stage 1: number analyzed (Participants) | 45 | 40 | 45 | 11
  Boys: Baseline-Stage 1 | 0 | 0 | 0 | 0
  Boys: Baseline-Stage 2: number analyzed (Participants) | 45 | 40 | 45 | 11
  Boys: Baseline-Stage 2 | 4 | 3 | 0 | 0
  Boys: Baseline-Stage 3: number analyzed (Participants) | 45 | 40 | 45 | 11
  Boys: Baseline-Stage 3 | 7 | 5 | 5 | 3
  Boys: Baseline-Stage 4: number analyzed (Participants) | 45 | 40 | 45 | 11
  Boys: Baseline-Stage 4 | 14 | 21 | 16 | 7
  Boys: Baseline-Stage 5: number analyzed (Participants) | 45 | 40 | 45 | 11
  Boys: Baseline-Stage 5 | 20 | 11 | 24 | 1
  Boys: Month 24-Stage 1: number analyzed (Participants) | 29 | 28 | 24 | 6
  Boys: Month 24-Stage 1 | 0 | 0 | 0 | 0
  Boys: Month 24-Stage 2: number analyzed (Participants) | 29 | 28 | 24 | 6
  Boys: Month 24-Stage 2 | 0 | 0 | 0 | 0
  Boys: Month 24-Stage 3: number analyzed (Participants) | 29 | 28 | 24 | 6
  Boys: Month 24-Stage 3 | 2 | 2 | 1 | 0
  Boys: Month 24-Stage 4: number analyzed (Participants) | 29 | 28 | 24 | 6
  Boys: Month 24-Stage 4 | 9 | 13 | 8 | 2
  Boys: Month 24-Stage 5: number analyzed (Participants) | 29 | 28 | 24 | 6
  Boys: Month 24-Stage 5 | 18 | 13 | 15 | 4
  Girls: Baseline-Stage 1: number analyzed (Participants) | 53 | 49 | 42 | 9
  Girls: Baseline-Stage 1 | 0 | 0 | 0 | 0
  Girls: Baseline-Stage 2: number analyzed (Participants) | 53 | 49 | 42 | 9
  Girls: Baseline-Stage 2 | 0 | 1 | 0 | 0
  Girls: Baseline-Stage 3: number analyzed (Participants) | 53 | 49 | 42 | 9
  Girls: Baseline-Stage 3 | 8 | 3 | 6 | 1
  Girls: Baseline-Stage 4: number analyzed (Participants) | 53 | 49 | 42 | 9
  Girls: Baseline-Stage 4 | 17 | 21 | 16 | 8
  Girls: Baseline-Stage 5: number analyzed (Participants) | 53 | 49 | 42 | 9
  Girls: Baseline-Stage 5 | 28 | 24 | 20 | 0
  Girls: Month 24- Stage 1: number analyzed (Participants) | 27 | 30 | 27 | 5
  Girls: Month 24- Stage 1 | 0 | 0 | 0 | 0
  Girls: Month 24-Stage 2: number analyzed (Participants) | 27 | 30 | 27 | 5
  Girls: Month 24-Stage 2 | 0 | 0 | 0 | 0
  Girls: Month 24-Stage 3: number analyzed (Participants) | 27 | 30 | 27 | 5
  Girls: Month 24-Stage 3 | 0 | 0 | 0 | 0
  Girls: Month 24-Stage 4: number analyzed (Participants) | 27 | 30 | 27 | 5
  Girls: Month 24-Stage 4 | 5 | 9 | 9 | 1
  Girls: Month 24-Stage 5: number analyzed (Participants) | 27 | 30 | 27 | 5
  Girls: Month 24-Stage 5 | 22 | 21 | 18 | 4

31. Other Pre Specified Outcome: Time to Discontinuation Due to AEs
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Reporting Status: Not Posted

32. Secondary Outcome: Change From Baseline in the PANSS Total Score
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) to 7 (extremely severe symptoms). The PANSS total score was the sum of the rating scores for 7 positive scale items, 7 negative scale items, and 16 general psychopathology scale items from the PANSS panel. The PANSS total score ranges from 30 (best possible outcome) to 210 (worst possible outcome). Higher scores indicate worsening of symptoms. A negative change from baseline reflects improvement or reduction in symptom severity.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: Efficacy Sample consists of all participants in the Safety Sample who had a baseline assessment and at least one post-baseline assessment of the PANSS Total Score. The data for this outcome measure was planned to be collected for only OLT period arm groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 96 | 87 | 85 | 20
score on a scale | -18.44 (17.53) | -20.14 (17.63) | -19.76 (18.88) | -19.00 (13.61)

33. Secondary Outcome: Change From Baseline in the PANSS Positive Subscale Scores
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) to 7 (extremely severe symptoms). The PANSS total score was the sum of the rating scores for 7 positive (+ve) scale items, 7 negative (-ve) scale items, and 16 general psychopathology scale items from the PANSS panel. The PANSS total score ranges from 30 (best possible outcome) to 210 (worst possible outcome). Higher scores indicate worsening of symptoms. A negative change from baseline reflects improvement or reduction in symptom severity.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 96 | 87 | 85 | 20
score on a scale | -4.59 (5.11) | -5.20 (5.08) | -5.29 (5.75) | -5.15 (4.97)

34. Secondary Outcome: Change From Baseline in the PANSS Negative Subscale Scores
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) to 7 (extremely severe symptoms). The PANSS total score was the sum of the rating scores for 7 positive scale items, 7 negative scale items, and 16 general psychopathology scale items from the PANSS panel. The PANSS total score ranges from 30 (best possible outcome) to 210 (worst possible outcome). Higher scores indicate worsening of symptoms. A negative (-ve) change from baseline reflects improvement or reduction in symptom severity.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period)
Number analyzed (Participants) | 96 | 87 | 85 | 20
score on a scale | -4.82 (5.46) | -4.89 (4.98) | -4.55 (5.37) | -4.40 (4.11)

35. Secondary Outcome: Change From Baseline in Children's Global Assessment Scale (CGAS) Total Score
Description: The CGAS is a 100-point rating scale measuring psychological, social and school functioning for children aged 6-17. The scale is separated into 10-point sections with the score ranging from 0-100, 1 to 10 indicates the need for constant supervision and 91 to 100 indicates superior functioning in all areas. A positive change from baseline reflects improvement in functioning.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Prior Aripiprazole (Open-label Treatment Period): Participants who received aripiprazole in the previous study were administered brexpiprazole tablets, starting with a dose of 0.5 mg/day by Day 4, titrated up to 1 mg/day by Day 7, with a 1 mg increase or decrease if needed and tolerated, 1 or 2 mg/day by Days 14, 1-3 mg/ day by Days 21, up to a maximum dose of 4 mg by Day 22 in the current study
- Prior Placebo (Open-label Treatment Period): Participants who received brexpiprazole or aripiprazole matching placebo tablets in the previous study were administered brexpiprazole tablets, starting with a dose of 0.5 mg/day by Day 4, titrated up to 1 mg/day by Day 7, with a 1 mg increase or decrease if needed and tolerated, 1 or 2 mg/day by Days 14, 1-3 mg/ day by Days 21, up to a maximum dose of 4 mg by Day 22 in the current study
- De Novo (Open-label Treatment Period): De novo participants who rolled over from the previous study, and newly enrolled participants in this study were administered brexpiprazole tablets, starting with a dose of 0.5 mg/day by Day 4, titrated up to 1 mg/day by Day 7, with a 1 mg increase or decrease if needed and tolerated, 1 or 2 mg/day by Days 14, 1-3 mg/ day by Days 21, up to a maximum dose of 4 mg by Day 22. De novo participants, for whom a washout period was not appropriate in the opinion of the investigator entered a conversion period to cross-titrate from their current antipsychotic treatments to monotherapy with brexpiprazole 1, 2, or 3 mg/day and washout from prohibited medications. Participants who completed the conversion period entered the de novo open-label treatment period.
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole (Open-label Treatment Period) | Prior Placebo (Open-label Treatment Period) | De Novo (Open-label Treatment Period)
Number analyzed (Participants) | 96 | 87 | 85 | 20
score on a scale | 13.58 (13.26) | 14.31 (14.13) | 12.92 (13.42) | 23.05 (12.80)

36. Secondary Outcome: Mean Clinical Global Impression Severity (CGI-S) Scale Score
Description: The CGI-S scale is an investigator-rated evaluation that assesses the severity of a participant's illness on a 7-point scale, ranging from 1 to 7. The investigator answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" Response choices include: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients. Higher scores indicate worse condition.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole (Open-label Treatment Period) | Prior Placebo (Open-label Treatment Period) | De Novo (Open-label Treatment Period)
Number analyzed (Participants) | 96 | 87 | 85 | 20
score on a scale | -1.09 (1.16) | -1.11 (1.20) | -0.86 (1.21) | -1.30 (1.08)

37. Secondary Outcome: Mean Clinical Global Impression - Improvement (CGI-I) Scale Score
Description: The efficacy of brexpiprazole in the treatment was rated for each participant using the CGI-I. The investigator rated the participant's total improvement whether or not it was entirely due to drug treatment on a 7-point scale, ranging from 0 to 7. Response choices were: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. Higher scores indicate worse condition.
Time Frame: From the first dose of the study drug up to the last dose in the open-label treatment period (Up to Month 24)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior & Current Brexpiprazole (OLT Period) | Prior Aripiprazole (Open-label Treatment Period) | Prior Placebo (Open-label Treatment Period) | De Novo (Open-label Treatment Period)
Number analyzed (Participants) | 96 | 87 | 85 | 20
score on a scale | 2.1 (1.2) | 2.1 (1.1) | 2.2 (1.1) | 1.9 (1.1)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug (including the open-label treatment period and the conversion period in the current study) up to 21 days after the last dose of study drug (up to approximately 25.6 months)
Description: The safety population included all enrolled participants who received at least one dose of the study drug. Participants with conversion were analyzed separately in addition to their analysis in treatment period arms.
Groups:
- Prior and Current Brexpiprazole: Participants who received brexpiprazole in the previous study 331-10-234 were administered brexpiprazole tablets, orally, once a day (QD) at a starting dose of 0.5 mg/day from Day 1 to Day 4 in this study. Thereafter, the dose was titrated to 1 mg/day by Day 7, with the option of a 1 mg increase or decrease if needed and tolerated. The dose was adjusted within the range of 1 mg/day to 2 mg/day by Day 14, 1 mg/day to 3 mg/ day by Day 21, and up to a maximum of 4 mg/day by Day 22 based on clinical judgement. Participants continued to receive flexible dose of brexpiprazole (1 mg/day to 4 mg/day) up to Month 24. Participants were followed for safety for another 21 days. Open-label Treatment Period = OLT Period.
- Prior Aripiprazole & Current Brexpiprazole (OLT Period): Participants who received aripiprazole in the previous study 331-10-234, were administered brexpiprazole tablets, orally, QD at a starting dose of 0.5 mg/day from Day 1 to Day 4 in this study. Thereafter, the dose was titrated to 1 mg/day by Day 7, with the option of a 1 mg increase or decrease if needed and tolerated. The dose was adjusted within the range of 1 mg/day to 2 mg/day by Day 14, 1 mg/day to 3 mg/ day by Day 21, and up to a maximum of 4 mg/day by Day 22 based on clinical judgement. Participants continued to receive flexible dose of brexpiprazole (1 mg/day to 4 mg/day) up to Month 24. Participants were followed for safety for another 21 days.
- Prior Placebo & Current Brexpiprazole (OLT Period): Participants who received brexpiprazole or aripiprazole matching placebo tablets in the previous study 331-10-234, were administered brexpiprazole tablets, orally, QD at a starting dose of 0.5 mg/day from Day 1 to Day 4 in this study. Thereafter, the dose was titrated to 1 mg/day by Day 7, with the option of a 1 mg increase or decrease if needed and tolerated. The dose was adjusted within the range of 1 mg/day to 2 mg/day by Day 14, 1 mg/day to 3 mg/ day by Day 21, and up to a maximum of 4 mg/day by Day 22 based on clinical judgement. Participants continued to receive flexible dose of brexpiprazole (1 mg/day to 4 mg/day) up to Month 24. Participants were followed for safety for another 21 days.
- De Novo (OLT Period): De novo participants who rolled over from the previous study 331-10-234, and newly enrolled participants in this study were administered brexpiprazole tablets, orally, QD, at a starting dose of 0.5 mg/day from Day 1 to Day 4. Thereafter, the dose was titrated to 1 mg/day by Day 7, with the option of a 1 mg increase or decrease if needed and tolerated. The dose was adjusted within the range of 1 mg/day to 2 mg/day by Day 14, 1 mg/day to 3 mg/ day by Day 21, and up to a maximum of 4 mg/day by Day 22 based on clinical judgement. Participants continued to receive flexible dose of brexpiprazole (1 mg/day to 4 mg/day) up to Month 24. Participants were followed for safety for another 21 days.
- De Novo (Conversion Period): Participants underwent a cross-titration to oral brexpiprazole 1, 2, or 3 mg/day for 1 to 4 weeks to achieve the required washout of prohibited medications during the conversion period.
Arm/Group | Prior and Current Brexpiprazole | Prior Aripiprazole & Current Brexpiprazole (OLT Period) | Prior Placebo & Current Brexpiprazole (OLT Period) | De Novo (OLT Period) | De Novo (Conversion Period)
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/89 | 0/87 | 0/20 | 0/14
Serious Adverse Events (participants affected / at risk) | 4/98 | 1/89 | 3/87 | 1/20 | 0/14
Other Adverse Events (participants affected / at risk) | 45/98 | 37/89 | 42/87 | 13/20 | 5/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior and Current Brexpiprazole (N=98) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) (N=89) | Prior Placebo & Current Brexpiprazole (OLT Period) (N=87) | De Novo (OLT Period) (N=20) | De Novo (Conversion Period) (N=14)
Abnormal Sensation in Eye (Eye disorders) | 1 | 0 | 0 | 0 | 0
Pilonidal Disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Psychomotor Hyperactivity (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior and Current Brexpiprazole (N=98) | Prior Aripiprazole & Current Brexpiprazole (OLT Period) (N=89) | Prior Placebo & Current Brexpiprazole (OLT Period) (N=87) | De Novo (OLT Period) (N=20) | De Novo (Conversion Period) (N=14)
Erythropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Hyperprolactinaemia (Endocrine disorders) | 0 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 3 | 1 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 1 | 0
Coronavirus Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 4 | 5 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 9 | 6 | 4 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 2 | 5 | 0 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Coronavirus Test Positive (Investigations) | 0 | 0 | 0 | 2 | 0
Weight Increased (Investigations) | 7 | 12 | 9 | 4 | 0
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 2 | 0
Akathisia (Nervous system disorders) | 6 | 4 | 4 | 1 | 1
Headache (Nervous system disorders) | 10 | 9 | 11 | 0 | 0
Sedation (Nervous system disorders) | 1 | 2 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 9 | 7 | 9 | 6 | 2
Tension Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 4 | 4 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 4 | 8 | 1 | 1
Intentional Self-Injury (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Major Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Emotional Disorders (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Initial Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT03238326/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT03238326/SAP_001.pdf